CLINICAL TRIAL: NCT00660140
Title: A Phase II Study of Gemcitabine and Carboplatin in the Treatment of Metastatic or Recurrent Cholangiocarcinoma/Gallbladder Cancer
Brief Title: Study of Gemcitabine and Carboplatin in the Treatment of Metastatic or Recurrent Cholangiocarcinoma/Gallbladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-0925
Record Dates: First submitted 2008-04-11; First posted 2008-04-17 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Cholangiocarcinoma; Gallbladder Cancer
Keywords: Cholangiocarcinoma; Gallbladder; Cancer
MeSH Terms: conditions — Cholangiocarcinoma; Gallbladder Neoplasms; Neoplasms | interventions — Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine + Carboplatin (Experimental): Gemcitabine 1000 mg/m2 IV for 30 minutes on days 1 and 8 of 21 day cycle. Maximum of 9 cycles.
  Carboplatin AUC 5 IV for 1 hour on day 1 of 21 day cycle. Maximum of 9 cycles.
  Interventions: Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Gemcitabine
  Other Names: Gemzar
Drug: Carboplatin
  Other Names: Paraplatin; Paraplatin-AQ

SUMMARY:
To determine the activity of gemcitabine combined with carboplatin in the treatment of patients with metastatic or recurrent cholangiocarcinoma or gallbladder cancer.

DETAILED DESCRIPTION:
Due to better non-hematologic toxicity profile, less need for pre- and post chemotherapy hydration, and tolerability as compared to cisplatin, we propose to combine gemcitabine with carboplatin in the treatment of patients with cholangiocarcinoma and gallbladder carcinoma. In lung cancer, available literature suggests that carboplatin is as efficacious as cisplatin.

Several Phase I, II and III studies using gemcitabine with carboplatin have already been done or are currently ongoing. Phase I studies determined the maximum tolerated doses (MTD) of gemcitabine at 800-1250 mg/m2 days 1 and 8 combined with at AUC of 4-5.5, day 1 of a 21-day cycle.

Initial Phase II studies using a 28-day schedule using gemcitabine on days 1,8 and 15 with carboplatin caused severe thrombocytopenia on day 15 precluding day 15 treatment in over 50% of courses. A Spanish Lung Cancer Group conducted a sequential Phase II trial wherein 52% and 30% of the first 33 patients with lung cancer treated using the 28-day schedule were noted to have Grade 4 thrombocytopenia and neutropenia, respectively. Subsequently, the next 56 patients were treated on the 21-day schedule, and despite a higher dose intensity, response rates were equal (45-48%) with less Grade 4 thrombocytopenia (21%) but similar rates of Grade 4 neutropenia (27%).

A randomized Italian Phase II studies have demonstrated that when gemcitabine was given at doses of 1 g/m2 with carboplatin at AUC of 5 mg/mL/min were tolerable and when compared to gemcitabine and cisplatin caused less non-hematologic toxicities. Current Phase III trials in lung cancer utilizes the 21-day schedule with gemcitabine at 1000 mg/m2 on days 1 and 8 and carboplatin at AUC of 5.5.

Therefore, our proposed schedule will be gemcitabine at 1000 mg/m2 IV over 30 minutes on days 1 and 8 with carboplatin dosed at an AUC of 5 on day 1 of a 21-day cycle.

ELIGIBILITY:
1. Patients must have biopsy-proven locally-advanced, metastatic or recurrent adenocarcinoma of the biliary ducts or gallbladder.
2. Patients must have measurable disease.
3. Patients must be 18 years or older.
4. Patients must have a NCI CTC Performance Status of 0-2.
5. Patients must have a life expectancy of >= 3 months.
6. Patients must not have any prior chemotherapy for metastatic disease. Prior adjuvant radiation therapy and chemotherapy with 5FU and/or gemcitabine is allowed.
7. At least 3 weeks should have elapsed since any surgery requiring general anesthesia.
8. Patients must have no prior malignancies except for basal or squamous skin cancers, cervical carcinoma-in-situ.
9. Pregnant patients are not eligible. Non-pregnant status will be determined in all women of childbearing potential. All patients will be required to use an effective means of contraception if sexually active during therapy.
10. Initial Required Laboratory Values:

    * 1. Absolute neutrophil count >= 1,500/mm3, platelet count >= 100,000/mm3, and hemoglobin >= 9 g/dL.
    * 2. Serum creatinine should be <= 2 mg/dL.
    * 3. Serum bilirubin should be <= 3.0 mg/dL (biliary stents allowed).
    * 4. Serum transaminases should be <= 5-fold the institutional upper limits.
11. Patients must not have any co-existing severe medical illnesses, such as unstable angina, uncontrolled diabetes mellitus, uncontrolled arrhythmia or uncontrolled infection.
12. Patients must be able to sign an informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2002-03; Primary Completion 2007-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To determine the response rate and time to failure for patients treated with this regimen | Every 3 cycles for a maximum of 9 cycles
  1 cycle = 21 days

SECONDARY OUTCOMES:
To describe the toxicities associated with gemcitabine and carboplatin in patients with cholangiocarcinoma or gallbladder cancer. | 30 days after last dose of study drug
To assess the clinical benefit, or lack thereof, of chemotherapy on patient's performance status and weight. | At the end of study treatment
Time to progression | Every 3 months until progression
Survival times | Every 3 months until patient death

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Tan, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Williams KJ, Picus J, Trinkhaus K, Fournier CC, Suresh R, James JS, Tan BR. Gemcitabine with carboplatin for advanced biliary tract cancers: a phase II single institution study. HPB (Oxford). 2010 Aug;12(6):418-26. doi: 10.1111/j.1477-2574.2010.00197.x. PMID 20662793
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu